CLINICAL TRIAL: NCT03070262
Title: Caffeic Acid for Advanced Esophageal Squamous Cell Cancer: A Randomized, Double-blind, and Multicenter Trial in Chinese Patients
Brief Title: The Efficacy and Safety of Caffeic Acid for Esophageal Cancer
Acronym: CAEC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital of Henan University of Science and Technology (Other)
Collaborators: Anyang Tumor Hospital (Other); 150th Hospital of PLA (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GiCAEC-LY001
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-04

CONDITIONS: Esophagus Cancer
Keywords: esophageal cancer; caffeic acid
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CA group (Experimental): caffeic acid (300mg, tid, po) continue given until progression of disease or death, or patients are unable to bear the side effects
  Interventions: Drug: CA
- placebo group (Placebo Comparator): the same shape placebo tablets continue given until progression of disease or death, or patients are unable to bear the side effects
  Interventions: Drug: placebo group

INTERVENTIONS:
Drug: CA — caffeic acid, 300mg, tid, po
  Arms: CA group
Drug: placebo group — placebo tablet, 3 tablets, tid, po
  Arms: placebo group

SUMMARY:
Caffeic acid can target inhibit GASC1 (gene amplified in squamous cell carcinoma 1, also known as KDM4C and JMJD2C) expression and GASC1 is confirmed to be a new oncogene in several cancers including esophageal cancer. This study aims to investigate the efficiency and safety of coffeic acid in chinese advanced esophageal squamous cell cancer (ESCC).

DETAILED DESCRIPTION:
Background: More than half of global esophageal cancer cases came from China.80 percentage patients were diagnosed with advanced disease and suffered from the poor outcome.With the development of target therapy among cancers,the overall survival and life quality of patients has been continuous improved recently.However,there had little reports focusing on target therapy in esophageal cancer . Caffeic acid as an ordinary drug is used for thrombocytopenia when patient received chemotherapy. Newly studies shown caffeic acid can target inhibit GASC1 expression, and GASC1 is confirmed to be a new oncogene in esophageal cancer.

Aim: to investigate the efficiency and safety of caffeic acid in chinese advanced esophageal squamous cell cancer.

Methods: 240 advanced ESCC patients will be randomized to two arms: Arm A (receiving coffeic acid treatment) or Arm B (placebo group). In Arm A, patients will receive coffeic acid treatment: 300mg, tid, po, continue to progress disease (PD) or die or the intolerant adverse events; in Arm B, the same shape placebo tablets will be deliveried to patients. 1 years follow-up for both groups patients.Patients in both arms can receive any other ways of anti cancer therapy in the same time.

Primary endpoints: OS Second endpoints: PFS

ELIGIBILITY:
Inclusion Criteria:

* Chinese
* esophageal squamous cell cancer
* stage IV or disease recurrence
* chemotherapy, or radiotherapy, or palliative care is going on

Exclusion Criteria:

* PS (performance status): ≥ 3
* severe hepatic and renal dysfunction
* hypercoagulability
* thrombocytosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | 1 year
  The percentage of 1 year overall survival (OS) after random allocation. The follow-up will be done every 3 months through phone call, investigator visiting, and medical recording review.

SECONDARY OUTCOMES:
progression-free survival (PFS) | 1 year
  The percentage of 3 months progression-free survival (PFS) after random allocation. PFS was defined as the time from randomisation to disease progression or death as assessed by the treating physicians in the study through CT scan, gastroscopy and biopsy pathology, X-ray barium meal.

CONTACTS AND LOCATIONS:
Overall Officials: Shegan Gao, PhD, Study Chair — The Clinical Medical College, The First Affiliated Hospital of Henan Science and Technology
Locations (1):
- The Clinical Medical College, The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li S, Zhang W, Yang Y, Ma T, Guo J, Wang S, Yu W, Kong L. Discovery of oral-available resveratrol-caffeic acid based hybrids inhibiting acetylated and phosphorylated STAT3 protein. Eur J Med Chem. 2016 Nov 29;124:1006-1018. doi: 10.1016/j.ejmech.2016.10.028. Epub 2016 Oct 15. PMID 27783972
- [Result] Pedersen MT, Kooistra SM, Radzisheuskaya A, Laugesen A, Johansen JV, Hayward DG, Nilsson J, Agger K, Helin K. Continual removal of H3K9 promoter methylation by Jmjd2 demethylases is vital for ESC self-renewal and early development. EMBO J. 2016 Jul 15;35(14):1550-64. doi: 10.15252/embj.201593317. Epub 2016 Jun 6. PMID 27266524
- [Result] Movassaghian S, Xie Y, Hildebrandt C, Rosati R, Li Y, Kim NH, Conti DS, da Rocha SR, Yang ZQ, Merkel OM. Post-Transcriptional Regulation of the GASC1 Oncogene with Active Tumor-Targeted siRNA-Nanoparticles. Mol Pharm. 2016 Aug 1;13(8):2605-21. doi: 10.1021/acs.molpharmaceut.5b00948. Epub 2016 Jun 27. PMID 27223606
- [Result] Sudo G, Kagawa T, Kokubu Y, Inazawa J, Taga T. Increase in GFAP-positive astrocytes in histone demethylase GASC1/KDM4C/JMJD2C hypomorphic mutant mice. Genes Cells. 2016 Mar;21(3):218-25. doi: 10.1111/gtc.12331. Epub 2016 Jan 25. PMID 26805559
- [Result] Ye Q, Holowatyj A, Wu J, Liu H, Zhang L, Suzuki T, Yang ZQ. Genetic alterations of KDM4 subfamily and therapeutic effect of novel demethylase inhibitor in breast cancer. Am J Cancer Res. 2015 Mar 15;5(4):1519-30. eCollection 2015. PMID 26101715
- [Result] Ozaki Y, Fujiwara K, Ikeda M, Ozaki T, Terui T, Soma M, Inazawa J, Nagase H. The oncogenic role of GASC1 in chemically induced mouse skin cancer. Mamm Genome. 2015 Dec;26(11-12):591-7. doi: 10.1007/s00335-015-9592-9. Epub 2015 Aug 7. PMID 26248577
- [Result] Sun LL, Wu JY, Wu ZY, Shen JH, Xu XE, Chen B, Wang SH, Li EM, Xu LY. A three-gene signature and clinical outcome in esophageal squamous cell carcinoma. Int J Cancer. 2015 Mar 15;136(6):E569-77. doi: 10.1002/ijc.29211. Epub 2014 Sep 24. PMID 25220908
- [Result] Uimonen K, Merikallio H, Paakko P, Harju T, Mannermaa A, Palvimo J, Kosma VM, Soini Y. GASC1 expression in lung carcinoma is associated with smoking and prognosis of squamous cell carcinoma. Histol Histopathol. 2014 Jun;29(6):797-804. doi: 10.14670/HH-29.797. Epub 2013 Dec 27. PMID 24371038
- [Result] Sun LL, Holowatyj A, Xu XE, Wu JY, Wu ZY, Shen JH, Wang SH, Li EM, Yang ZQ, Xu LY. Histone demethylase GASC1, a potential prognostic and predictive marker in esophageal squamous cell carcinoma. Am J Cancer Res. 2013 Nov 1;3(5):509-17. eCollection 2013. PMID 24224128
- [Result] Berdel B, Nieminen K, Soini Y, Tengstrom M, Malinen M, Kosma VM, Palvimo JJ, Mannermaa A. Histone demethylase GASC1--a potential prognostic and predictive marker in invasive breast cancer. BMC Cancer. 2012 Nov 14;12:516. doi: 10.1186/1471-2407-12-516. PMID 23148692
- [Result] Liu G, Bollig-Fischer A, Kreike B, van de Vijver MJ, Abrams J, Ethier SP, Yang ZQ. Genomic amplification and oncogenic properties of the GASC1 histone demethylase gene in breast cancer. Oncogene. 2009 Dec 17;28(50):4491-500. doi: 10.1038/onc.2009.297. Epub 2009 Sep 28. PMID 19784073
- [Result] Yuan X, Kong J, Ma Z, Li N, Jia R, Liu Y, Zhou F, Zhan Q, Liu G, Gao S. KDM4C, a H3K9me3 Histone Demethylase, is Involved in the Maintenance of Human ESCC-Initiating Cells by Epigenetically Enhancing SOX2 Expression. Neoplasia. 2016 Oct;18(10):594-609. doi: 10.1016/j.neo.2016.08.005. Epub 2016 Sep 19. PMID 27742014
- [Result] Tyszka-Czochara M, Konieczny P, Majka M. Caffeic Acid Expands Anti-Tumor Effect of Metformin in Human Metastatic Cervical Carcinoma HTB-34 Cells: Implications of AMPK Activation and Impairment of Fatty Acids De Novo Biosynthesis. Int J Mol Sci. 2017 Feb 21;18(2):462. doi: 10.3390/ijms18020462. PMID 28230778
- [Result] Bonuccelli G, De Francesco EM, de Boer R, Tanowitz HB, Lisanti MP. NADH autofluorescence, a new metabolic biomarker for cancer stem cells: Identification of Vitamin C and CAPE as natural products targeting "stemness". Oncotarget. 2017 Mar 28;8(13):20667-20678. doi: 10.18632/oncotarget.15400. PMID 28223550
- [Result] Chung LC, Chiang KC, Feng TH, Chang KS, Chuang ST, Chen YJ, Tsui KH, Lee JC, Juang HH. Caffeic acid phenethyl ester upregulates N-myc downstream regulated gene 1 via ERK pathway to inhibit human oral cancer cell growth in vitro and in vivo. Mol Nutr Food Res. 2017 Sep;61(9). doi: 10.1002/mnfr.201600842. Epub 2017 Mar 20. PMID 28181403
- [Result] Dziedzic A, Kubina R, Kabala-Dzik A, Tanasiewicz M. Induction of Cell Cycle Arrest and Apoptotic Response of Head and Neck Squamous Carcinoma Cells (Detroit 562) by Caffeic Acid and Caffeic Acid Phenethyl Ester Derivative. Evid Based Complement Alternat Med. 2017;2017:6793456. doi: 10.1155/2017/6793456. Epub 2017 Jan 12. PMID 28167973
- [Result] Sirota R, Gibson D, Kohen R. The timing of caffeic acid treatment with cisplatin determines sensitization or resistance of ovarian carcinoma cell lines. Redox Biol. 2017 Apr;11:170-175. doi: 10.1016/j.redox.2016.12.006. Epub 2016 Dec 7. PMID 27951496